CLINICAL TRIAL: NCT04160182
Title: Feasibility and Effectiveness of an Internet-based Intervention to Manage Fatigue in Breast Cancer Survivors
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID this trial never got up and running.
Sponsor: University of Toledo Health Science Campus (Other)
Collaborators: University of Toledo (Other)
Responsible Party: Sponsor
Organization: University of Toledo (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UT BCS ECS Study
Record Dates: First submitted 2019-11-01; First posted 2019-11-12 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer; Fatigue
Keywords: Breast cancer; fatigue; Intervention
MeSH Terms: conditions — Breast Neoplasms; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Energy Conservation Work Simplification Education (Experimental): The intervention will be delivered online by an occupational therapist. The intervention consists of 6 weekly sessions; each session will be 45 minutes long. The focus of the intervention is to teach breast cancer survivors strategies to manage their fatigue.
  Interventions: Behavioral: Energy Conservation Work Simplification Education

INTERVENTIONS:
Behavioral: Energy Conservation Work Simplification Education — The intervention will last approximately 45 minutes, and will be provided once/week for 6 weeks. The intervention is delivered "live" using web-cameras (e.g., Microsoft Zoom).
  Registered and licensed occupational therapists will deliver the intervention. At beginning of the intervention, the participant and interventionist prioritize the 5 most critical fatigue-related problems that they would like to solve during the intervention. Each week, the interventionist will guide the participant through a workbook to provide knowledge and examples on how to apply the knowledge to everyday fatigue-related problems. The workbook contains: (a) information regarding fatigue in breast cancer survivors, (b) knowledge regarding fatigue management strategies, and (c) worksheets to develop skills to recognize and solve fatigue-related problems. Participants will retain the workbook after study completion.

SUMMARY:
The purpose of this project is to determine the feasibility and effectiveness of a 6-week, internet-based, Energy Conservation and Activity Management intervention among women who report cancer-related fatigue following breast cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer diagnoses
* not currently receiving active treatment in the form of chemotherapy or radiation therapy
* at least 18 years of age
* fatigue severe enough to limit daily activities (score ≥ 4 on 7-point Fatigue Severity Scale)(Krupp, LaRocca, Muir-Nash, & Steinberg, 1989);
* functional English fluency and literacy;
* Participant has a smart device that operates on the Android or Apple platform
* Participant is able to use the Ecological Momentary Assessment application before going to bed every night

Exclusion Criteria:

* self-reported history of diagnosis of co-morbidities that have been associated with poor sleep and fatigue: chronic insomnia, chronic fatigue syndrome, unstable heart, lung, or neuromuscular disease, insulin-dependent diabetes, sleep apnea, chronic oral steroid therapy, and night-shift employment,
* Disability due to a diagnosis other then breast cancer
* Currently taking medication for depression, sleep issues, or fatigue.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-27 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Change in Fatigue Scores (Revised Piper Fatigue Scale) | Baseline to 14 weeks
  Measure of fatigue severity and impact

SECONDARY OUTCOMES:
Change in Fatigue Impact (Patient Reported Outcomes Measurement Information System Fatigue Scale) | Baseline to 14 weeks
  Measure of fatigue severity and impact
Change in Fatigue Impact (Modified Fatigue Impact Scale) | Baseline at 14 weeks
  Measure of fatigue impact
Change in Severity of Fatigue Measured Via Ecological Momentary Assessments | Baseline to 14 weeks
  Ecological Momentary Assessments via Smartphone App

CONTACTS AND LOCATIONS:
Overall Officials: Ketki Raina, PhD, OTR/L, Principal Investigator — University of Toledo
Locations (1):
- University of Toledo, Toledo, Ohio, United States

IPD SHARING:
Plan to Share IPD: No